CLINICAL TRIAL: NCT02322749
Title: A Phase I, Single Centre, Randomised, Open Label, Crossover Study to Assess the Bioequivalence or Relative Bioavailability of Variants of Selumetinib (AZD6244, Hyd-Sulfate) Blue Capsules in Healthy Male Volunteers Aged 18 to 45 Years
Brief Title: A Study to Assess the Relative Bioavailability of Process Variants of Selumetinib in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00078
Record Dates: First submitted 2014-12-09; First posted 2014-12-23 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers Bioequivalence or Bioavailability Study
Keywords: bioequivalence; bioavailability; pharmacokinetics; Phase I; AZD6244; cancer
MeSH Terms: conditions — Neoplasms | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): AZD6244 blue reference capsules (3 x 25 mg) administered orally
  Interventions: Drug: selumetinib 75mg single dose
- Treatment B (Experimental): AZD6244 blue capsules (3 x 25 mg) Variant 1 (free base variant) administered orally
  Interventions: Drug: selumetinib 75mg single dose
- Treatment C (Experimental): AZD6244 blue capsules (3 x 25 mg) Variant 2 (vitamin E polyethylene glycol succinate [TPGS] variant) administered orally
  Interventions: Drug: selumetinib 75mg single dose

INTERVENTIONS:
Drug: selumetinib 75mg single dose — 3 blue capsules of 25 mg given as a single dose
  Other Names: Selumetinib
  Arms: Treatment A
Drug: selumetinib 75mg single dose — 3 capsules of 25 mg given as a single dose
  Other Names: Selumetinib
  Arms: Treatment B
Drug: selumetinib 75mg single dose — 3 capsules of 25 mg given as a single dose
  Other Names: Selumetinib
  Arms: Treatment C

SUMMARY:
A Study to assess, against a reference selumetinib capsule, if the drug levels of a variant of selumetinib capsule are comparable, and to assess how drug levels differed in another variant of Selumetinib in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:1.Provision of written informed consent 2.Healthy male volunteers aged 18 to 45 years 3.Calculated creatinine clearance (CrCL) >50 mL/minute using the Cockcroft-Gault formula 4.Healthy volunteers with sexual partners who could become pregnant should agree to use 2 highly effective methods of contraception. Healthy volunteers with sexual partners who are pregnant should agree to use an effective method of contraception (barrier method) from the first administration until 12 weeks after the last administration of the investigational product. Healthy volunteers should avoid sperm donation during the study and for 12 weeks after the last administration of the investigational product 5.Use no nicotine containing products for at least 3 months prior to screening 6.For inclusion in the genetic component of the study, healthy volunteers provide written informed consent for genetic research.

Exclusion Criteria:

1.Healthy male volunteers of Japanese or non Japanese Asian, or Indian ethnicity 2.Any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian or Indian 3.Involvement in the planning and/or conduct of the study. 4.Previous randomisation to treatment in the present study 5.Participation in another clinical study within 3 month before Visit 1, or participation in a method development study 1 month before Visit 1. 6.Current or past history of central serous retinopathy or retinal vein thrombosis, intraocular pressure greater than 21 mmHg or uncontrolled glaucoma 7.Any clinically significant disease or disorder that may put the healthy volunteer at risk because of participation in the study, influence the result of the study or influence the healthy volunteer's ability to participate in the study 8.Any clinically relevant abnormal findings in physical examination, haematology, clinical chemistry, urinalysis, vital signs or 12-lead ECG at Visit 1, which may put the healthy volunteer at risk because of his participation in the study. 9.Use of prescribed medications and over-the-counter drugs (including herbal remedies) known to have moderate or strong cytochrome P450 (CYP) 3A4 or CYP2C19 inducer or inhibitory effects from 30 days prior to the first administration of investigational product until the follow up visit 10.Use of any other prescribed medications and over-the-counter drugs (including herbal remedies, vitamins and minerals) within 2 weeks or 5 times the half life, whichever is longer, of the respective drug prior to Visit 2, with the exception of occasional use of acetaminophen (paracetamol or TYLENOL®) and over-the-counter adrenergic nasal spray for relief of nasal congestion. No medications known to prolong the QT/corrected QT interval (QTc) interval are allowed 11.Excessive intake of caffeine containing drinks or food. 12.Any intake of grapefruit and Seville oranges or other products containing grapefruit or Seville oranges within 7 days of the first admission 13.A definite or suspected personal history of intolerance or hypersensitivity to drugs and/or their excipients 14.Plasma donation or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening 15.History of, or current alcohol or drug abuse. 16.A suspected/manifested infection according to the International Air Transport Association (IATA) Categories A and B infectious substances 17.Healthy male volunteers who do not agree to use at least 2 effective methods of contraception 18.Positive results at screening for human immunodeficiency virus (HIV) and/or hepatitis B and/or hepatitis C 19.Planned inpatient surgery, dental procedure or hospitalisation during the study 20.Healthy male volunteers who, in the opinion of the Principal Investigator, should not participate in the study 21.Healthy male volunteers with a LVEF <55% 22.Previous bone marrow transplant 23.Whole blood transfusion within 120 days of the genetic sample collection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olufeyikemi Oluwayi, MBChB, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 healthy adult males were enrolled in this single centre, randomised, open label, 3-period, 3-treatment and 6-sequence crossover study from 24 February 2015 to study completion on 30 April 2015. Subjects attended the clinical study unit for at least 1 screening visit and 3 treatment periods.
Pre-assignment Details: 48 subjects received at least 1 of the 3 treatments and 45 completed all 3 treatment periods. There was a washout period of 7 to 10 days between administrations. A follow-up visit occurred 7 days after the last administration of the third treatment period.
Groups:
- Sequence ABC: Subjects randomized to treatment sequences ABC: A=Selumetinib Blue Reference Capsules; B=Selumetinib Blue Free Base Variant Capsules; C=Selumetinib Blue TPGS Variant Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
- Sequence ACB: Subjects randomized to treatment sequences ACB: A=Selumetinib Blue Reference Capsules; C=Selumetinib Blue TPGS Variant Capsules; B=Selumetinib Blue Free Base Variant Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
- Sequence BAC: Subjects randomized to treatment sequences BAC: B=Selumetinib Blue Free Base Variant Capsules; A=Selumetinib Blue Reference Capsules; C=Selumetinib Blue TPGS Variant Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
- Sequence BCA: Subjects randomized to treatment sequences BCA: B=Selumetinib Blue Free Base Variant Capsules; C=Selumetinib Blue TPGS Variant Capsules; A=Selumetinib Blue Reference Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
- Sequence CAB: Subjects randomized to treatment sequences CAB: C=Selumetinib Blue TPGS Variant Capsules; A=Selumetinib Blue Reference Capsules; B=Selumetinib Blue Free Base Variant Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
- Sequence CBA: Subjects randomized to treatment sequences CBA: C=Selumetinib Blue TPGS Variant Capsules; B=Selumetinib Blue Free Base Variant Capsules; A=Selumetinib Blue Reference Capsules. Subjects received 75 mg selumetinib (3 x 25 mg capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration) in a crossover fashion. There was a washout period of 7-10 days between administrations.
Period: Period 1
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 6 | 8 | 8
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 8 | 8 | 8 | 6 | 8 | 8
Completed | 8 | 8 | 7 | 6 | 8 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects (n = 48) were included in the baseline analysis
Groups:
- Overall Study: All subjects received at least 1 dose of selumetinib. Subjects were randomised in a crossover fashion to receive 1 of 3 treatments during each treatment period: Period 1=Visit 2; Period 2=Visit 3; Period 3=Visit 4.
Arm/Group | Overall Study
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence of the Free Base Variant of Selumetinib (Treatment B) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib Cmax]
Description: The bioequivalence of the free base variant of selumetinib (Treatment B) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the maximum observed plasma concentration (Cmax) of selumetinib in healthy volunteers.
Time Frame: Blood samples were collected pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post dose for each of the separate treatment periods (Visits 2, 3 and 4).
Population: The Pharmacokinetic (PK) analysis set included all healthy subjects who received at least 1 dose of selumetinib and had at least 1 post-dose PK measurement without important protocol deviations/violations or events significantly affecting the PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Groups:
- Treatment A: Selumetinib Blue Reference Capsules: Subjects received 75 mg selumetinib (3 x 25 mg blue reference capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration).
- Treatment B: Selumetinib Blue Free Base Variant Capsules: Subjects received 75 mg selumetinib (3 x 25 mg free base variant capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration).
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules
Number analyzed (Participants) | 46 | 48
nanograms per millilitre (ng/mL) | 1330 (36.6) | 124 (50.3)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment B: Selumetinib Blue Free Base Variant Capsules; Test type: Non-Inferiority or Equivalence — If the 90% confidence intervals for both AUC and Cmax were entirely contained within the limits 80.00% to 125.00% then bioequivalence was concluded; Geometric Least Squares (LS) Mean Ratio = 9.32, 90% CI 2-sided [8.25 to 10.53] — Selumetinib: Ratio of Treatment B to Treatment A based on a linear mixed-effects model with sequence, period, and treatment as fixed effects and volunteer nested within sequence as a random effect

2. Primary Outcome: Bioequivalence of the Free Base Variant of Selumetinib (Treatment B) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib AUC]
Description: The bioequivalence of the free base variant of selumetinib (Treatment B) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC) of selumetinib in healthy volunteers.
Time Frame: as for outcome 1
Population: The PK analysis set included all healthy subjects who received at least 1 dose of selumetinib and had at least 1 post-dose PK measurement without important protocol deviations/violations or events significantly affecting the PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * hour per mL (ng*h/mL)
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules
Number analyzed (Participants) | 45 | 41
ng * hour per mL (ng*h/mL) | 3750 (24.1) | 905 (32.6)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment B: Selumetinib Blue Free Base Variant Capsules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 24.26, 90% CI 2-sided [22.62 to 26.03] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Bioequivalence of the Free Base Variant of Selumetinib (Treatment B) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib AUC(0-t)]
Description: The bioequivalence of the free base variant of selumetinib (Treatment B) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the AUC from time zero to the time of the last quantifiable concentration (AUC[0-t]) of selumetinib in healthy volunteers.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules
Number analyzed (Participants) | 45 | 48
ng*h/mL | 3670 (24.0) | 814 (32.2)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment B: Selumetinib Blue Free Base Variant Capsules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS mean ratio = 22.12, 90% CI 2-sided [20.65 to 23.69] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Relative Bioavailability of the TPGS Capsule Variant (Treatment C) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib Cmax]
Description: The relative bioavailability of the TPGS capsule variant of selumetinib (Treatment C) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the Cmax of selumetinib in healthy volunteers.
Time Frame: Blood samples were collected pre-dose, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose for each of the separate treatment periods (Visits 2, 3 and 4).
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment C: Selumetinib Blue TPGS Variant Capsules: Subjects received 75 mg selumetinib (3 x 25 mg vitamin E polyethylene glycol succinate [TPGS] variant capsules) administered as a single oral dose on Day 1 of each period according to their treatment sequence under fasted conditions (10 hours prior to administration).
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Number analyzed (Participants) | 46 | 44
ng/mL | 1330 (36.6) | 172 (46.5)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment C: Selumetinib Blue TPGS Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 12.93, 90% CI 2-sided [11.42 to 14.65] — Selumetinib: Ratio of Treatment C to Treatment A based on a linear mixed-effects model with sequence, period, and treatment as fixed effects and volunteer nested within sequence as a random effect

5. Secondary Outcome: Relative Bioavailability of the TPGS Capsule Variant (Treatment C) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib AUC]
Description: The relative bioavailability of the TPGS capsules variant of selumetinib (Treatment C) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the AUC of selumetinib in healthy volunteers.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Number analyzed (Participants) | 45 | 40
ng*h/mL | 3750 (24.1) | 975 (31.7)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment C: Selumetinib Blue TPGS Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 26.20, 90% CI 2-sided [24.44 to 28.09] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Relative Bioavailability of the TPGS Capsule Variant (Treatment C) Compared to the Blue Reference Capsule (Treatment A) [Selumetinib AUC(0-t)]
Description: The relative bioavailability of the TPGS capsule variant of selumetinib (Treatment C) as compared to the blue reference capsule (Treatment A) was evaluated by comparing the AUC[0-t] of selumetinib in healthy volunteers.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Number analyzed (Participants) | 45 | 44
ng*h/mL | 3670 (24.0) | 866 (31.4)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment C: Selumetinib Blue TPGS Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 23.60, 90% CI 2-sided [22.02 to 25.30] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: The PK of the Metabolite N-desmethyl Selumetinib by Assessment of Cmax
Description: The PK of the metabolite N-desmethyl selumetinib was evaluated by assessing the Cmax of the metabolite in healthy volunteers after oral administration of single doses of the blue reference capsule (Treatment A), the free base variant capsule (Treatment B) and the TPGS variant capsule (Treatment C).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Number analyzed (Participants) | 46 | 48 | 44
ng/mL | 95.2 (34.8) | 9.13 (50.9) | 12.3 (48.6)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment B: Selumetinib Blue Free Base Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 9.66, 90% CI 2-sided [8.5 to 10.97] — N-desmethyl selumetinib: Ratio of Treatment B to Treatment A based on a linear mixed-effects model with sequence, period, and treatment as fixed effects and volunteer nested within sequence as a random effect
Statistical Analysis 2: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment C: Selumetinib Blue TPGS Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 13.04, 90% CI 2-sided [11.45 to 14.86] — N-desmethyl selumetinib: Ratio of Treatment C to Treatment A based on a linear mixed-effects model with sequence, period, and treatment as fixed effects and volunteer nested within sequence as a random effect

8. Secondary Outcome: The PK of N-desmethyl Selumetinib by Assessment of the AUC(0-t)
Description: The PK of the metabolite N-desmethyl selumetinib was evaluated by assessing the AUC(0-t) of the metabolite in healthy volunteers after oral administration of single doses of the blue reference capsule (Treatment A), the free base variant capsule (Treatment B) and the TPGS variant capsule (Treatment C).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Number analyzed (Participants) | 45 | 48 | 44
ng*h/mL | 267 (31.1) | 30.2 (72.1) | 33.9 (66.2)
Statistical Analysis 1: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment B: Selumetinib Blue Free Base Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 11.31, 90% CI 2-sided [9.80 to 13.05] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Treatment A: Selumetinib Blue Reference Capsules vs Treatment C: Selumetinib Blue TPGS Variant Capsules; Test type: Superiority or Other; Geometric LS Mean Ratio = 12.80, 90% CI 2-sided [11.07 to 14.80] — [estimate comment as in outcome 7, analysis 2]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from randomisation (Visit 2, Day 1) until the follow-up visit (Visit 5).
Description: Visits 2, 3 and 4 comprised 3 separate treatment periods with a washout period of 7 - 10 days between administrations.
Arm/Group | Treatment A: Selumetinib Blue Reference Capsules | Treatment B: Selumetinib Blue Free Base Variant Capsules | Treatment C: Selumetinib Blue TPGS Variant Capsules
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 12/46 | 12/48 | 9/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Selumetinib Blue Reference Capsules (N=46) | Treatment B: Selumetinib Blue Free Base Variant Capsules (N=48) | Treatment C: Selumetinib Blue TPGS Variant Capsules (N=45)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter Site Related Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 6 (7) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Party (PI or Sponsor) will use the other Party's name in connection with any publication or promotion without the other Party's prior, written consent.